CLINICAL TRIAL: NCT03851237
Title: Novel CCR2 PET for Pancreatic Cancer Imaging and Prediction of Response to Standard and CCR2-Targeted Therapy
Brief Title: CCR2 PET for Pancreatic Cancer Imaging and Prediction of Response to Standard and CCR2-Targeted Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201807099; 1R01CA235672-01 (NIH)
Record Dates: First submitted 2019-02-14; First posted 2019-02-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1a: Treatment Whipple/Surgical Procedure/Surgery following neoadjuvant therapy (Experimental): * Early-staged localized pancreatic cancer
  * Standard of care diagnostic biopsy
  * 64Cu-DOTA-ECL1i-PET/CT imaging - immediately after the dynamic study
  * Receive treatment with upfront surgery such as whipple procedure or surgery following neoadjuvant therapy.
- Cohort 1b: Standard of Care Treatment Chemotherapy (Experimental): * Borderline resectable, locally advanced/metastatic or recurrent pancreatic cancer
  * Standard of care diagnostic biopsy (if available tissue to be used for CCR2 expression)
  * 64Cu-DOTA-ECL1i-PET/CT imaging pretherapy
  * Treatment with any standard of care (SOC) chemotherapy
  * Additional 64Cu-DOTA-ECL1i-PET/CT imaging for patients with positive scan at baseline/early therapy at the time of standard of care follow-up imaging appointment --Additional 64Cu-DOTA-ECL1i-PET/CT imaging for patients with negative scan at baseline/early therapy at time recurrence is diagnosed by any standard imaging modality
  Interventions: Drug: 64Cu-DOTA-ECLIi; Device: PET/CT
- Cohort 2: CCR2-Targeted Therapy (Experimental): * Locally advanced or borderline resectable pancreatic cancer
  * Biopsy per therapeutic protocol (if available tissue to be used for CCR2 expression)
  * 64Cu-DOTA-ECL1i-PET/CT imaging pretherapy
  * 2 cycles of CCR2-targeted therapy
  * Biopsy per therapeutic protocol (tissue to be used for CCR2 expression) --Additional 64Cu-DOTA-ECL1i-PET/CT imaging after 2 cycles of therapy
  Interventions: Drug: 64Cu-DOTA-ECLIi; Device: PET/CT

INTERVENTIONS:
Drug: 64Cu-DOTA-ECLIi — -The first four patients enrolled on study will undergo an additional delayed imaging time point approximately 2-6 hours following 64Cu-DOTA-ECL1i
  Arms: Cohort 1b: Standard of Care Treatment Chemotherapy; Cohort 2: CCR2-Targeted Therapy
Device: PET/CT — -Standard of care
  Arms: Cohort 1b: Standard of Care Treatment Chemotherapy; Cohort 2: CCR2-Targeted Therapy

SUMMARY:
Currently there is no clinical biomarker that can be used to select patients for CCR2-targeted therapy and to monitor response to such therapy. Considering the toxicity and the rate of response to CCR2-targeted therapy, it is crucial to be able to identify patients who may not response to this therapy in order to avoid the morbidity and expense associated with ineffective therapy.

Therefore, the combination of the novel CCR2 imaging agent with the novel CCR2-targeted therapy in this trial is of great importance to promote science while prolonging the life and its quality in patients with PDAC. The investigators also believe that this combination will make substantial contributions to the fields of cancer immunotherapy and tumor monocyte/macrophage biology. Moreover, this imaging agent has the potential to not only facilitate development and testing of future CCR2-targeted therapeutic agents but also serve as a prescreen tool to select appropriate patients for imaging guided treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age or older with:

  * newly diagnosed early-staged localized pancreatic ductal adenocarcinoma (PDAC) scheduled to undergo Whipple procedure (cohort 1a) or down-staged after neoadjuvant chemotherapy now eligible to undergo resection OR
  * borderline resectable, locally advanced, metastatic, or recurrent PDAC (cohort 1b) scheduled to undergo chemotherapy OR
  * borderline resectable, locally advanced PDAC (cohort 2) who is eligible and / or signed consent to undergo CCR2-targeted therapy example:[(phase 1/2 clinical trial combining an oral CCR2/5i (BMS-813160) with chemotherapy (gemcitabine plus nab-paclitaxel) and anti-PD-1 (nivolumab), PI, Dr. Kian Lim) HRPO #201806007 - closed to accrual March 2022] AND
  * at least one measurable [defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan or MRI] A cohort 1B subject who has been previously treated for PDAC with a diagnosis of recurrence and a lesion size of 1.5 cm or greater will be allowed to enroll before institution of therapy or within 20 days after starting a 2nd line or later (new therapy) for recurrent disease.
* Able to give informed consent
* Not currently pregnant or nursing: Subject must be surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), post-menopausal (cessation of menses for more than 1 year), non-lactating, or of childbearing potential for whom a urine pregnancy test (with the test performed within the 24 hour period immediately prior to administration of 64Cu-DOTA-ECL1i) is negative

Exclusion Criteria:

* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of the other cancer present within the last 5 years
* Unable to tolerate up to 90 min of PET/CT imaging per imaging session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Determine whether 64Cu-DOTA-ECL1i detects CCR2 expression in PDAC tumors as measured by direct comparison of visual tumor uptake on 64Cu-DOTA-ECL1i images to CCR2 measurements in surgical specimens | At any of the following time points: prior to the start of any chemotherapy or change in chemotherapy, pre-surgery without intervention or pre-surgery with intervention
  * Visual tumor uptake as compared to background blood/tissue uptake: 1=no uptake, 2=mild uptake, 3=moderate uptake, and 5=striking update
  * Will utilize published methods of immunohistochemical staining techniques
Evaluate whether tumor uptake of 64Cu-DOTA-ECL1i prior to therapy (systemic therapy or surgery) or following neoadjuvant therapy prior to surgery predicts response to standard of care chemotherapy as measured by tumor SUVmax | Completion of first scan (day 1)
  SUVmax is a mathematical measurement of tumor burden seen on images and calculated by the following equation SUVmax= r / (a'/w) where r= radioactivity concentration in tumor (kBq/ml) as measured by the PET scanner within a defined region of interest, a'=the decay corrected amount of injected 64Cu-DOTA-ECL1i and w= weight of the patient in grams When PET imaging shows uptake of 64Cu-DOTA-ECL1i in site(s) of known tumor the SUVmax will be compared to clinical measurement of response to treatment taking into consideration standard response criteria including radiological imaging, laboratory values, physical examination and repeat pathology as applicable.
Evaluate whether tumor take of 64Cu-DOTA-ECL1i post therapy correlates with CCR2 expression and is predictive of response to therapy as measured by visual tumor uptake on 64Cu-DOTA-ECL1i images | Baseline and after 2 cycles of CCR directed therapy (estimated to be 2 months)
  * Visual tumor uptake as compared to background blood/tissue uptake: 1=no uptake, 2=mild uptake, 3=moderate uptake, and 5=striking update
  * A decrease in visual tumor uptake from baseline to post therapy imaging in cohort 2 subject is hypothesized to represent response to CCR2 directed therapy while an increase in tumor uptake is expected in cohort 1b subjects who progress while receiving standard therapy.
Evaluate if tumor take of 64Cu-DOTA-ECL1i is predictive of response to CCR2-directed therapy measured by comparison of SUVmax at imaging prior to the start of CCR2 directed therapy and SUVmax at imaging performed after 2 cycles of CCR2 directed therapy | Baseline and after 2 cycles of CCR2 directed therapy (estimated to be 2 months)
  * Cohort 2 only
  * SUVmax is a mathematical measurement of tumor burden seen on images and calculated by the following equation SUVmax= r / (a'/w) where r= radioactivity concentration in tumor (kBq/ml) as measured by the PET scanner within a defined region of interest, a'=the decay corrected amount of injected 64Cu-DOTA-ECL1i and w= weight of the patient in grams When PET imaging shows uptake of 64Cu-DOTA-ECL1i in site(s) of known tumor the SUVmax will be evaluated for change at baseline and after 2 cycles of CCR2 directed therapy. SUVmax measurements will also be compared to clinical measurement of response to treatment taking into consideration standard response criteria including radiological imaging, laboratory values, physical examination and repeat pathology as applicable

CONTACTS AND LOCATIONS:
Overall Officials: Farrokh Dehdashti, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu